CLINICAL TRIAL: NCT03127306
Title: Validation of the Polish Version of the Behavioral Pain Scale in a Postoperative Cardiac Surgery Unit.
Brief Title: Validation of the Polish Version of BPS (POL-BPS).
Acronym: POL-BPS
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Katarzyna Kotfis, Katarzyna Kotfis M.D. Ph.D., Pomeranian Medical University Szczecin
Other Study IDs: POL-BPS
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Pain, Acute
Keywords: Pain; Behavioural Pain Scale; BPS; NRS; Delirium; CAM-ICU
MeSH Terms: conditions — Acute Pain; Pain; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CAM-ICU (+) Delirious patients.: Behavioral: BPS assessment
  Polish version of BPS tool validation.
  Other Names:
  Pain assessment in non-verbal patients
  Interventions: Diagnostic Test: Assessment of Polish version of BPS
- CAM-ICU (-) Non-delirious patients.: Behavioral: BPS assessment
  Polish version of BPS tool validation.
  Other Names:
  Pain assessment in non-verbal patients
  Interventions: Diagnostic Test: Assessment of Polish version of BPS

INTERVENTIONS:
Diagnostic Test: Assessment of Polish version of BPS — Validation of Polish Version of BPS.

SUMMARY:
Between 40 to 70% of patients with critical illness experience moderate to severe pain. Diagnosing pain and assessing its severity is difficult in non-verbal patients both in an Intensive Care Unit and in Postoperative Unit after a major surgery such as cardiac surgery). In patients who are unable to self-report pain, we use behavioural pain scales, namely BPS - Behavioural Pain Scale.

Aim: The aim of this study was to validate the Polish version of a behavioural pain assessment method - BPS in intubated, sedated patients after cardiac surgery versus self assessment of pain using Numeric rating scale (NRS) in both delirious and non-delirious patients (assessed using Confusion Assessment Method for ICU, CAM-ICU).

Method: A prospective observational cohort study will include 60 patients. The patients will be observed by two trained observers during a nociceptive procedure (position change), both during analgosedation and analgesia. Patients will be observed 5 minutes before, during, and 15 min after the two sets of interventions (six assessments in total). Each BPS assessment will be carried out by two observers blinded to each other. To validate the Polish BPS translation we will use the following methods: calculations of interrater reliability, criterion validity and discriminant validity.

DETAILED DESCRIPTION:
Patients after major surgery, namely cardiac surgery frequently suffer pain during their postoperative stay in the intensive care unit. Nearly 30% of those patients experience pain at rest and up to 50% experience pain during nursing procedures. Pain experienced by critically ill patients falls into four categories that coexist and overlap: pre-existing chronic pain, acute illness-related pain, continuous ICU treatment-related pain or discomfort and intermittent procedural pain. Moreover, acute pain experienced in the ICU may become a chronic problem after discharge from the unit, as a lifelong ICU footprint. Everyday nursing procedures, including position changing performed in the ICU may be a potential source of pain, therefore there is a clinical need for a simple and easy behavioural pain scale to evaluate this condition in patients unable to self assess pain.

Assessment of pain in patients treated in the ICU becomes a daily clinical challenge for the ICU team, also in those units where minimal sedation environment based on analgesia are used. Various guidelines and recommendations exist to guide the ICU care team in the pain management and assessment process. Nevertheless, the gold standard for pain assessment is patient's self-report of pain (using numeric raing scale - NRS), which can be aided with behavioural scales only when the self-report is unreliable or impossible to obtain. Observational pain scales include the Behavioural Pain Scale (BPS) and have been recommended for clinical use in the critically ill adults. However, their validation in a given patient population (cardiac, burn, different languages) is strongly recommended and required.

The need to equip critical care teams (intensive care units - ICUs, high dependency unit - HDUs, Post-Operative Units) with dedicated monitoring tools is clear. The BPS has been developed by critical care professionals and validated in various situations, but it has not been translated or validated in Polish until now.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Ability to communicate in the Polish language,
* Intubated and mechanically ventilated patients (controlled modes, spontaneous modes),
* Richmond Agitation Sedation Scale (RASS) above or equal to -3,
* Unrestricted sight and hearing,
* No limitations for body position changing,
* After Cardiac surgery

Exclusion Criteria:

* A medical need for deep sedation - treatment of severe respiratory failure associated with patient-ventilator dyssynchrony, preventing awareness during neuromuscular blockade, status epilepticus, certain surgical conditions requiring immobility , cases of severe brain injury with intracranial hypertension
* Facial trauma (unable to evaluate facial expression),
* Richmond Agitation Sedation Scale (RASS) -4 or -5
* Neurological or psychiatric disorders,
* Use of neuromuscular blocking agents,
* Regular narcotic users,
* Chronic pain syndrome patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intubated adult ICU patients at the Postoperative Cardiac Surgery Unit of the tertiary teaching hospital at the Pomeranian Medical University in Szczecin, Poland undergoing minimal analgesia-based sedation protocol (dexmedetomidine + morphine intravenous infusion).
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Interrater variability for Polish BPS. | Through study completion and up to 24 weeks.
  Validation of Polish BPS.

SECONDARY OUTCOMES:
Criterion validity for Polish BPS. | Through study completion and up to 24 weeks.
  Validation od Polish BPS.
Discriminant validity for Polish BPS | Through study completion and up to 24 weeks.
  Validation of Polish BPS.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna L Kotfis, MD,PhD, Principal Investigator — Pomeranian Medical University
Locations (1):
- Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: Undecided